CLINICAL TRIAL: NCT03510312
Title: Long-term Prognosis in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji Hoe Heo, Professor, Severance Hospital
Other Study IDs: 4-2011-0731
Record Dates: First submitted 2016-12-28; First posted 2018-04-27 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Long-term follow up, observational: This cohort does not involve interventions, just follow up of prognosis of ischemic stroke/transient ischemic attack patients.

SUMMARY:
A single-center cohort of patients with acute ischemic stroke and transient ischemic attack who admitted to the Severance hospital of Yonsei university and their long-term outcomes.

DETAILED DESCRIPTION:
This is a single-center cohort of consecutive patients with acute ischemic stroke and transient ischemic attack who admitted to the Severance hospital of Yonsei university in Republic of Korea.

Stroke recurrence, Cardiovascular event, all cause mortality and cardiovascular mortality were collected through long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute ischemic stroke or transient ischemic attack

Exclusion Criteria:

* A patient who did not agree with enrollment of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with acute ischemic stroke/transient ischemic attack
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2011-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Event of Stroke or transient ischemic attack | through study completion, up to 10 years
  The time of a stroke or transient ischemic attack occurs (through study completion)
Event of cardiovascular disease (include stroke/transient ischemic attack) | through study completion, up to 10 years
  The time of a cardiovascular disease (stroke/transient ischemic attack) occurs (through study completion)
All cause mortality | through study completion, up to 10 years
  The time of death from any cause (through study completion)
Cardiovascular cause mortality (include stroke/transient ischemic attack mortality) | through study completion, up to 10 years
  The time of death from cardiovascular cause (through study completion)
The modified Rankin Scale (mRS) | 3 months
  Measure functional outcome as the form of mRS at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoe Heo, MD, PhD, Study Chair — Yonsei University
Locations (1):
- Ji Hoe Heo, Seoul, South Korea